CLINICAL TRIAL: NCT05541991
Title: Randomized, Double-blind, Placebo-controlled Clinical Study Evaluating the Effect of Rhubarb Extract Supplementation on Stool Frequency and Biological Markers of Intestinal Function in Seniors With a Low Number of Defecations Per Week
Brief Title: Study on the Effect of Rhubarb Extract on Stool Frequency and Biological Markers of Intestinal Function in Seniors With Low Defecation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ortis (Industry)
Collaborators: CEN Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C1486
Record Dates: First submitted 2022-08-24; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Constipation - Functional

STUDY DESIGN:
Intervention Model Description: Randomized double-blind clinical study versus placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single dose product (Experimental): A single dose coated tablet with standardised rhubarb extract is administrated daily in the evening during 30days
  Interventions: Dietary Supplement: single dose coated tablet Fruits & Fibres Rhubarbe with standardised rhubarb extract
- Double dose product (Experimental): A double dose coated tablet with standardised rhubarb extract is administrated daily in the evening during 30days
  Interventions: Dietary Supplement: double dose coated tablet Fruits & Fibres Rhubarbe with standardised rhubarb extract
- placebo product (Placebo Comparator): A placebo coated tablet without active is administrated daily in the evening during 30days
  Interventions: Dietary Supplement: placebo coated tablet

INTERVENTIONS:
Dietary Supplement: single dose coated tablet Fruits & Fibres Rhubarbe with standardised rhubarb extract — coated tablet with a single dose of standardised rhubarb extract
  Arms: Single dose product
Dietary Supplement: placebo coated tablet — coated tablet without active principle
  Arms: placebo product
Dietary Supplement: double dose coated tablet Fruits & Fibres Rhubarbe with standardised rhubarb extract — coated tablet with a double dose of standardised rhubarb extract
  Arms: Double dose product

SUMMARY:
Randomized double-blind clinical study versus placebo evaluating the effect of supplementation with rhubarb extract on stool frequency and biological markers of intestinal function in seniors with a low number of defecations per week

DETAILED DESCRIPTION:
The main objective was to evaluate the effect of rhubarb extract supplementation on improving intestinal transit in subjects with a low number of defecations per week.

The secondary objectives are to assess: changes in the appearance of the stool; the evolution of the quality of life; the evolution of biological markers of intestinal function; the evolution of the intestinal microbiota; the evolution of low-grade chronic inflammatory markers; the evolution of endotoxemia; the evolution of oxidative stress; the relief experienced; subject satisfaction; the evolution of safety dosages; subject compliance.

The main efficacy criterion is the improvement in intestinal transit assessed by the frequency of stool emissions reported daily from D-14 to D 30.

The secondary endpoints correspond to the evolution of the aspect of the stools evaluated by the Bristol Stool Scale and the evolution of the quality of life evaluated by the SF-12.

They also correspond to the relief of the subjects evaluated on the PGII scale, to the tolerance of the product over the entire study period and in particular the occurrence of diarrhea and to the description of satisfaction on a Likert scale.

Regarding the biological assays, they correspond to:

* for biological markers of intestinal function to those specific to intestinal transit, i.e. active GLP-1, total GIP total PYY, PP (DPPIV substrates), Leptin, Insulin, by blood samples at D0 and D30 and that specific for permeability intestinal or claudin-3 by urine samples at D0 and D30;
* for the microbiota, analysis of bacterial taxa by PCR and metagenomics carried out on faecal samples collected on D0 and D30;
* for chronic low-grade chemokine inflammatory markers, Prostaglandins, interleukins, pro- and anti-inflammatory cytokines, ultra-sensitive CRP by blood samples at D0 and D30;
* for the measurement of endotoxaemia in the analysis of circulating LPS, TRL2 and 4 by blood samples on D0 and D30;
* for the measurement of oxidative stress to the ROS and NADPH oxidase content by blood serum samples at D0 and D30;
* for the safety assays for the lipid profile, NFS, glycaemia, kalemia, transaminases by blood samples on D0 and D30.

The studied product is a food supplement composed of a rhubarb extract standardized, characterized and optimized in order to improve these functional effects on the intestinal system (regulation of the local inflammatory system, microflora, peristalsis, etc.) at 2 different doses. The food supplement comes in the form of a film-coated tablet. The comparator product was a placebo with an appearance strictly identical to the verum and contains only excipients.

ELIGIBILITY:
Inclusion Criteria:

* presenting a number of stools ≥1 and ≤3 per week during the last month preceding the screening visit and during the last 15 days preceding the inclusion visit;
* stools often (at least 25% of defecations according to the Rome III questionnaire) hard or lumpy, according to the bristol scale, at least the last 3 months over a period of 6 months;
* not currently justifying, according to his attending physician, drug treatment;
* Giving free and informed consent to the study in writing.

Exclusion Criteria:

Related to the patient:

* subject with signs requiring further investigations: odynophagia, involuntary weight loss >10% during the last 3 months before inclusion, persistent vomiting, hematemesis, blood in the stools, iron deficiency anemia, symptoms of obstruction, rectal bleeding, rectal prolapse …;
* subject who has not been screened for colon cancer in the past two years;
* subject participating in another therapeutic trial;
* subject with a serious general pathology and in particular renal or hepatic insufficiency, cancer, chronic pancreatitis;
* premenopausal women;
* subject with known hypersensitivity to one of the constituents of the product under study;
* subject who does not have the legal or ethical capacity to contract due to an impairment of his cognitive functions;
* subject likely not to be compliant with the constraints imposed by the protocol;
* subject not benefiting from a health insurance scheme.

Related to the disorders assessed:

* subject having taken in the 30 days preceding the screening visit or currently taking medication, food supplements and any food enriched or presented as containing substances, bacteria or yeasts likely to have an effect on the intestines and more particularly on intestinal transit, digestive comfort, gas production, the occurrence of abdominal pain. These products were also prohibited throughout the duration of the study;
* subject following a particular diet (vegetarian, vegan, high protein, etc.);
* subject on a low-calorie diet and monitored by a current or recent doctor or dietitian (< 6 weeks);
* subject undergoing medical treatment which, according to the investigator, could interfere with the evaluation of the study criteria: antibiotic, corticosteroid, anticholinergic, antidepressant, antiemetic, antihistamine, diuretic, calcium channel blocker, antiparkinsonian, antipsychotic, antacid, analgesic , NSAIDs, H2 receptor antagonist, hypnotic, sedative, iron supplement, opioid and narcotic, laxative, anti-diarrheal, anti-reflux;
* subject with an alcohol consumption greater than 3 glasses of wine per day, or two pints of beer per day, or one glass of strong alcohol per day;
* subject with a coffee consumption greater than 5 cups per day;
* smoker;
* subject with a BMI greater than 30;
* subject with constipation attributable to an organic or anatomical cause (Hirschsprung's disease, hypothyroidism, mental deficiency, psychiatric illness, neurological abnormalities, history of colon or anus operation, colorectal cancer, anemia, etc.;
* subject with a fiber intake higher than the recommended intake (more than 6 fruits and vegetables per day according to the PNNS questionnaire);
* subject with severe constipation (less than 1 bowel movement per week during the 15 days preceding the inclusion visit);
* subject with pelvic floor dysfunction;
* subject with type 1 or 2 diabetes;
* subject with a history of pathology or current disorder at the gastrointestinal level such as a duodenal ulcer, chronic colitis or a chronic inflammatory disease of the digestive tract (Crohn's disease, ulcerative colitis), celiac disease or the syndrome irritable bowel;
* subject with a history of digestive tract surgery;
* subject having undergone surgery in the two months preceding the study;
* subject having undergone bariatric surgery;
* subject with the practice of an intense sports activity (more than 10 hours per week of intense activity as defined by the WHO).

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-06-13 (Actual)

PRIMARY OUTCOMES:
change of the number of defecations per week | Daily from Day -14 until the selection visit (Day 0) and every day during the 30days of treatment (until Day +30)
  The main objective was to evaluate the effect of rhubarb extract supplementation on changing intestinal transit in subjects with a low number of defecations per week.

SECONDARY OUTCOMES:
changes in the appearance of the stool | Daily from Day -14 until the selection visit (Day 0) and every day during the 30days of treatment (until Day +30)
  This secondary criteria correspond to the evolution of the aspect of the stools evaluated by the Bristol Stool Scale
the change of the quality of life | measured at Day -14 and Day +30 of the treatment
  the evolution of the quality of life is evaluated by the General quality of life score, not specific to a pathology (SF-12).
the evolution of biological markers of intestinal function | measured at Day 0 and Day +30 of the treatment
  for biological markers of intestinal function, this corresponds to those specific specific to intestinal permeability claudin-3 by urine samples at D0 and D30
the evolution of the biological marker of intestinal function, active GLP-1 | measured at Day 0 and Day +30 of the treatment
  for the biological marker of intestinal function: active GLP-1, this corresponds to those specific to intestinal transit, by blood samples at Day 0 and Day 30
the evolution of the biological marker of intestinal function, total GIP | measured at Day 0 and Day +30 of the treatment
  for the biological marker of intestinal function: total GIP, this corresponds to those specific to intestinal transit, by blood samples at Day 0 and Day 30
the evolution of the biological marker of intestinal function, total PYY | measured at Day 0 and Day +30 of the treatment
  for the biological marker of intestinal function: total PYY, this corresponds to those specific to intestinal transit, by blood samples at Day 0 and Day 30
the evolution of the biological marker of intestinal function, PP (DPPIV substrates) | measured at Day 0 and Day +30 of the treatment
  for the biological marker of intestinal function: PP (DPPIV substrates), this corresponds to those specific to intestinal transit, by blood samples at Day 0 and Day 30
the evolution of the biological marker of intestinal function, Leptin | measured at Day 0 and Day +30 of the treatment
  for the biological marker of intestinal function: total Leptin, this corresponds to those specific to intestinal transit, by blood samples at Day 0 and Day 30
the evolution of the biological marker of intestinal function, Insulin | measured at Day 0 and Day +30 of the treatment
  for the biological marker of intestinal function: total Insulin, this corresponds to those specific to intestinal transit, by blood samples at Day 0 and Day 30
the evolution of the intestinal microbiota by PCR | measured at Day 0 and Day +30 of the treatment
  for the microbiota, this corresponds to the analysis of bacterial taxa by PCR carried out on faecal samples collected on D0 and D30
the evolution of the intestinal microbiota by metagenomics | measured at Day 0 and Day +30 of the treatment
  for the microbiota, this corresponds to the analysis of bacterial taxa by metagenomics carried out on faecal samples collected on D0 and D30
the evolution of low-grade chronic inflammatory markers | measured at Day 0 and Day +30 of the treatment
  for low-grade chronic inflammatory markers, this corresponds to the dosage of chemokines, Prostaglandins, interleukins, pro- and anti-inflammatory cytokines, ultra-sensitive CRP by blood samples at D0 and D30
the evolution of endotoxemia | measured at Day 0 and Day +30 of the treatment
  for the measurement of endotoxemia, this corresponds to the analysis of circulating LPS, TRL2 and 4 by blood samples on D0 and D30
the evolution of oxidative stress | measured at Day 0 and Day +30 of the treatment
  for the measurement of oxidative stress, this corresponds to the ROS and NADPH oxidase content by blood serum samples at D0 and D30;
the relief experience | measured at Day +30 of the treatment
  It corresponds to the relief of the subjects evaluated on the Patient Global Impression of Improvement scale (PGII scale)
subject satisfaction | measured at Day +30 of the treatment
  It corresponds to the tolerance of the product over the entire study period and in particular the occurrence of diarrhea and to the description of satisfaction on a Likert scale.
the evolution of the incidence of treatment | measured at Day 0 and Day +30 of the treatment
  for the evolution of the incidence of treatment, this corresponds to the lipid profile, NFS, glycaemia, kalemia, transaminases by blood samples on D0 and D30.
subject compliance for taking the product | measured at Day +30 of the treatment
  Unused products are collected to assess compliance by measuring the number of unused product

CONTACTS AND LOCATIONS:
Overall Officials: Francois-andré Allaert, Principal Investigator — CEN Nutriment
Locations (1):
- CEN nutriment, Dijon, France

IPD SHARING:
Plan to Share IPD: No